CLINICAL TRIAL: NCT07350343
Title: The Predictability of Directly Printed Shape Memory (Graphy) Versus Thermoformed Clear Aligners: A Randomized Clinical Trial
Brief Title: The Predictability of Directly Printed Versus Thermoformed Clear Aligners
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hussin Anwar, Dentist.. PhD student, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1154425
Record Dates: First submitted 2026-01-05; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Class I Malocclusion; Crowded Teeth; Spacing of Anterior Teeth; Rotation
Keywords: direct printed graphy... thermoform
MeSH Terms: conditions — Malocclusion, Angle Class I; Crowding

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct-printed aligner (Graphy) (Experimental): Patients will be treated with direct-printed Graphy aligners until dental levelling alignment; space closure is finished.
  Interventions: Device: Direct-printed aligner (Graphy)
- Thermoformed aligner (Active Comparator): Patients will be treated with thermoformed aligners until dental alignment, levelling, space closure is finished.
  Interventions: Device: Thermoformed aligner

INTERVENTIONS:
Device: Direct-printed aligner (Graphy) — intraoral scanner would be used to scan patient teeth then aligner fabrication by direct printing then the patient will be treated with direct-printed aligners(graphy) until dental levelling alignment; space closure is finished. All patients would be given the same instructions: aligners had to be worn for at least 22 hours per day, except during meals and oral hygiene activities, and should be changed every 10 days.
  Arms: Direct-printed aligner (Graphy)
Device: Thermoformed aligner — intraoral scanner would be used to scan patient teeth then aligner fabrication by thermoforming then the Patients will be treated with thermoformed aligners (secret aligners) until dental alignment, levelling, space closure is finished. All patients would be given the same instructions: aligners had to be worn for at least 22 hours per day, except during meals and oral hygiene activities, and should be changed every 10 days.
  Arms: Thermoformed aligner

SUMMARY:
The study is randomized controlled trial ...The null hypothesis suggests that there is no significant difference between actual and predicted dental movement in patients treated using direct printed aligners produced with Graphy™ Tera Harz TA-28 resin as compared to those treated with thermoformed clear aligner therapy.

DETAILED DESCRIPTION:
the patients will be randomly assigned to one of two study groups which either direct printed or thermoformed clear aligner. All patients would be given the same instructions: aligners had to be worn for at least 22 hours per day, except during meals and oral hygiene activities, and should be changed every 10 days.Teeth positions would be planned according to esthetic and functional principles, starting with the 3D T0 digital model and aligning and leveling dental arches following orthodontic aligner biomechanical principles. Each aligner had a planned movement speed of 0.2 mm linear displacement, 2° long-axis rotation, and a vestibulo-lingual inclination of 2.5°.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate malocclusion that can be treated by less than 40 steps of aligner treatment, including those with dental rotation of < 30°, diastema or crowding of < 8 mm.
* Patients aged ≥ 16 years with fully erupted permanent teeth (regardless of the third molar).
* No supernumerary teeth, no enamel malformation.
* No tooth shape anomalies

Exclusion Criteria:

* Systemic pathologies such as uncontrolled diabetes or heart diseases
* active or past periodontal disease
* previous orthodontic treatment
* temporomandibular joint disorders
* ongoing pharmacological treatment could influence orthodontic treatment.

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
predictability of tooth movement | 12 months
  The primary outcome will be calculated as the percentage difference between the final and initial positions for each individual tooth movement assessed and will be expressed as a continuous numerical variable representing tooth movement predictability (%).

SECONDARY OUTCOMES:
predictability within different types | 12 months
  1. The secondary outcome will be assessed by comparing the predictability within different types of tooth movement of the same group.
Colour change of clear aligners | 12 months
  UV-Visible spectrophotometer for samples from both groups before and after intraoral aging.
Degree of Conversion | 12 months
  Assessment of the Degree of Conversion of direct printed Tera Harz TA-28 resin using Fourier-transform infrared (FTIR) spectroscopy for the liquid resin before curing and for samples after curing and post-processing.
shape memory effect | 12 months
  Assessment of the shape memory effect of direct printed Tera Harz TA-28 aligners, the bending test would be used to investigate and directly visualize the shape recovery property.

CONTACTS AND LOCATIONS:
Overall Officials: hussin anwar, Principal Investigator — University of Baghdad
Locations (1):
- The sample will be recruited from multicentre clinics (Private dental clinic, Orthodontic Department at Karbala Governmental Specialized Dental Centre, Orthodontic Department, College of Dentistry University of Baghdad)., Karbala, Iraq